CLINICAL TRIAL: NCT06702592
Title: Virtual Testicular Cancer Lay Support and Survivorship (VITALSS Study) Aim 2
Brief Title: Virtual Testis Cancer Lay Support and Survivorship Aim 2
Acronym: VITALSS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: LCCC2418 AIM2
Record Dates: First submitted 2024-11-20; First posted 2024-11-25 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Testicular Cancer; Testis Cancer
Keywords: virtual support; emotional well-being; self-efficacy; financial toxicity; quality of life
MeSH Terms: conditions — Testicular Neoplasms; Financial Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual support (Experimental): Participants will have access to the virtual support platform.
  Interventions: Behavioral: Virtual support
- Patient educational material (Other): Participants will have access to patient educational material only.
  Interventions: Behavioral: Patient educational material

INTERVENTIONS:
Behavioral: Virtual support — Subjects will use a virtual support platform that was built for their needs.
  Arms: Virtual support
Behavioral: Patient educational material — Participants will have access to patient educational material.
  Arms: Patient educational material

SUMMARY:
This study examines how virtual support can enhance well-being and survivorship in men with testicular cancer. Participants in North Carolina will be randomized into two groups: one with access to a virtual support platform and the other with access to patient educational materials only. After six months, the emotional well-being, self-efficacy, financial toxicity, and quality of life of both groups will be compared at 3 months and 6 months after baseline assessments.

ELIGIBILITY:
Inclusion Criteria:

* Men within 5 years of their initial diagnosis of germ cell testicular cancer.
* The subject is willing and able to comply with study procedures based on the judgment of the investigator.
* Adults aged 18-95 years old.
* Electronic informed consent was obtained to participate in the study.

Exclusion Criteria:

* Woman gender
* Non-English speaking
* Unwilling or unable to complete informed consent.
* On active treatment for another cancer.
* Actively receiving chemotherapy, radiation, or surgery for testicular cancer.

Ages: 18 Years to 95 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 360 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Emotional well-being scores comparison | At baseline, 3-months, and 6-months
  Emotional well-being will be assessed by patient-reported outcomes questionnaires using a 9-item Positive Affect and Well-Being assessment from the Neuro-QOL Item Bank v1. Emotional well-being scores in virtual support and enhanced usual care will be compared. It is a 5-point Likert scale, higher scores reflect better emotional well-being.

SECONDARY OUTCOMES:
Negative mental health comparison | At baseline, 3-months, and 6-months
  Negative mental health will be assessed by patient-reported outcomes questionnaires using 17 PROMIS items for anxiety, depression, loneliness, and stress. Negative mental health scores in virtual support and enhanced usual care will be compared. Scoring: Each item is rated on a 5-point scale between never (1) to always (5). The responses for each item are summed to get a total raw score. T-Scores: The raw score is then converted to a T-score using a scoring table specific to the PROMIS Anxiety item bank. T-scores standardize the results, making them comparable across different populations and studies. A T-score has a mean of 50 and a standard deviation of 10 in the general population.
Social well-being, acceptance and inclusion comparison | At baseline, 3-months, and 6-months
  Social well-being will be assessed by patient-reported outcomes questionnaires using the 6-item Acceptance/Inclusion subscale of the General Belongingness Scale (GBS). GBS measures an individual's sense of belonging and social connectedness. It consists of 12 items that assess feelings of acceptance and inclusion. Each item is rated on a 7-point Likert scale (1 = Strongly Disagree and 7 = Strongly Agree). Higher scores reflect better inclusion. Scores in virtual support and enhanced usual care will be compared.
Financial Toxicity comparison | At baseline, 3-months, and 6-months
  Financial Toxicity will be assessed by patient-reported outcomes questionnaires using a 12-item Comprehensive Score for Financial Toxicity (COST) instrument. Each item is rated on a 5-point Likert scale 0= = Not at all to 4= Very much. Higher scores indicate higher financial difficulties. Scores in virtual support and enhanced usual care will be compared.
Self-efficacy comparison | At baseline, 3-months, and 6-months
  Self-efficacy will be assessed by patient-reported outcomes questionnaires using 20 PROMIS items for self-efficacy for managing daily activities, emotions, social interactions, and symptoms. Self-efficacy scores in virtual support and enhanced usual care will be compared. Each item is rated on a 5-point scale ( 1 = Never, 5 = Always). Responses are summed to get a total raw score for each domain. Raw scores are converted to T-scores using a scoring table. T-scores standardize results, with a mean of 50 and a standard deviation of 10 in the general population.
Sexual Function and Satisfaction comparison | At baseline, 3-months, and 6-months
  Sexual Function and Satisfaction will be assessed by patient-reported outcomes questionnaires using a 20-item PROMIS SexFS instrument with domains for interest in sexual activity, global satisfaction with sex life, orgasm, and erectile function. Scores in virtual support and enhanced usual care will be compared. Each item is rated on a 5-point Likert scale: 1 = Not at all to 5= Very much. Raw scores are converted to T-scores using a scoring table specific to the PROMIS Sexual Function and Satisfaction profile. T-scores standardize the results, with a mean of 50 and a standard deviation of 10 in the general population.Higher T-scores indicate better sexual function and satisfaction.
Functional well-being comparison Functional well-being comparison | At baseline, 3-months, and 6-months
  Functional well-being will be assessed by patient-reported outcomes questionnaires using a 7-item subscale of the Functional Assessment of Cancer Therapy (FACT-G) instrument. Each item is rated on a 5-point Likert scale, 0= = Not at all to 4= Very much. Higher scores indicate better well-being. Scores in virtual support and enhanced usual care will be compared.
General Quality of Life comparison | At baseline, 3-months, and 6-months
  General Quality of Life will be assessed by patient-reported outcomes questionnaires using the PROMIS Global Health scale is an 8-item, validated survey that represents five core domains (physical function, pain, fatigue, emotional distress, social health). Two items each for physical and mental health as well as a question on quality of life will be administered. Scores in virtual support and enhanced usual care will be compared.
  Each item is rated on a 5-point Likert scale:1 = Poor to 5 = Excellent. Responses are summed to get a total raw score. The raw score is converted to a T-score using a scoring table. T-scores standardize the results, with a mean of 50 and a standard deviation of 10 in the general population. Higher T-scores indicate better overall health
General Self-Efficacy comparison | At baseline, 3-months, and 6-months
  General Self-Efficacy will be assessed by patient-reported outcomes questionnaires using the 4-item PROMIS instrument that measures the respondent's belief in managing specific problems or issues. Each item is scored on a 5-point Likert scale, 1 = Never to 5 = Always. The raw score is then converted to a T-score using a scoring table specific to the PROMIS domain being measured. T-scores standardize the results, with a mean of 50 and a standard deviation of 10 in the general population. Higher T-scores indicate more of the concept being measured Scores in virtual support and enhanced usual care will be compared.
Virtual platform usage | At baseline, 3-months, and 6-months
  Virtual platform usage will be assessed by time, visits, scrolling, posts, and messages spent on the virtual platform.
Healthcare and supportive care utilization | At baseline, 3-months, and 6-months
  Self-reported use of healthcare and supportive care services will be assessed by a survey. Participants will be asked to quantify healthcare or other supportive care visits over the intervention period.

CONTACTS AND LOCATIONS:
Overall Officials: Hung-Jui Tan, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clinical trials at UNC Lineberger — http://unclineberger.org/patientcare/clinical-trials/clinical-trials